CLINICAL TRIAL: NCT01585168
Title: Functional Neuroimaging of Alcoholism Vulnerability: Glutamate, Reward, Impulsivity and Pavlovian-to-Instrumental Transfer (PIT)
Brief Title: Functional Neuroimaging of Alcoholism Vulnerability (PIT)
Acronym: CTNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1106008650
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: Reward Circuitry; Impulsivity; Family History of Alcoholism; NMDA/DA Interactions
MeSH Terms: conditions — Impulsive Behavior | interventions — Memantine

STUDY DESIGN:
Intervention Model Description: All subjects received both the study drug and placebo. Family history was the main variable of interest, and randomization was stratified by this variable.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Family history positive, Memantine first, then placebo (Experimental): Memantine is a low-side-effect NMDA receptor antagonist usually administered therapeutically to elderly persons with moderately severe Alzheimer's disease in typical doses of 10-20 mg daily. In this study, single doses of 40 mg are administered.
  Interventions: Drug: Memantine; Drug: Placebo
- Family history positive, placebo first, then Memantine (Placebo Comparator): Memantine is a low-side-effect NMDA receptor antagonist usually administered therapeutically to elderly persons with moderately severe Alzheimer's disease in typical doses of 10-20 mg daily. In this study, single doses of 40 mg are administered.
  Interventions: Drug: Memantine; Drug: Placebo
- Family history negative, Memantine first, then placebo (Experimental): Memantine is a low-side-effect NMDA receptor antagonist usually administered therapeutically to elderly persons with moderately severe Alzheimer's disease in typical doses of 10-20 mg daily. In this study, single doses of 40 mg are administered.
  Interventions: Drug: Memantine; Drug: Placebo
- Family history negative, placebo first, then Memantine (Placebo Comparator): Memantine is a low-side-effect NMDA receptor antagonist usually administered therapeutically to elderly persons with moderately severe Alzheimer's disease in typical doses of 10-20 mg daily. In this study, single doses of 40 mg are administered.
  Interventions: Drug: Memantine; Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Memantine is a low-side-effect NMDA receptor antagonist usually administered therapeutically to elderly persons with moderately severe Alzheimer's disease in typical doses of 10-20 mg daily. In this study, single doses of 40 mg are administered.
Drug: Placebo — Identically appearing sugar pill, given orally

SUMMARY:
This project compares Family History Positive (FHP) for alcoholism subjects to matched Family History Negative (FHN) subjects derived from the project Principal Investigator's National Institute on Alcohol Abuse and Alcoholism-funded longitudinal study of drinking behavior in a 2000 college freshman population (known as the Brain and Alcohol Research in College Students study (BARCS)). The age of these subjects is a valuable one at which to capture the transition from harmful use to abuse/dependence. This project explores the effects of memantine in a double-blind, randomized, counterbalanced manner on alcoholism risk-relevant tasks. More specifically, this project studies functional MRI tasks related to different aspects of reward and/or impulsivity-related behavior in different contexts, compares the underlying neural circuitry across tasks, and uses a pharmacologic probe of the glutamatergic system to examine NMDA/DA interactions. The combined measures provide the opportunity to advance our understanding of specific aspects of brain function related to familial alcoholism vulnerability in an already well-characterized population as some members evolve into alcohol abuse. In addition to conventional within-task analyses, functional network connectivity and allied approaches will be used to examine brain networks across tasks.

The investigators will study adult male and female subjects in equal numbers who are either offspring of an alcoholic parent or are FHN matched controls. The investigators will recruit and assess a total of 84 (42 FHP and 42 matched FHN) subjects between the ages of 18-21 years on initial BARCS contact. The investigators will use 4 cognitive tasks during the functional MRI (fMRI) which include: 1) a Monetary Incentive Delay Task that distinguishes networks engaged in motivational (anticipation) and consummatory (outcome) components of reward processing; 2) a Go/No-Go Task that measures the ability to inhibit response to a pre-potent stimulus; 3) an Alcohol Cue Reactivity Task that examines Nucleus Accumbens response to alcohol-related versus matched soft drink stimuli; and 4) a Pavlovian-to-Instrumental Transfer (PIT) Task that dissects a component of the Monetary Incentive Delay (MID) Task, and provides an imaging assay of a transfer-like process that can be related to real-world drinking behavior, thus informing upon and extending the key findings from CTNA-2.

ELIGIBILITY:
Inclusion Criteria:

* Biological father with a history of Alcoholism
* A least 1 other first- or second-degree relative with a history of Alcoholism.

Exclusion Criteria:

* Cannot be an only child
* A diagnosis of DSM-IV-TR Axis I psychotic disorders screened with the Mini International Neuropsychiatric Interview (MINI), done in the BARCS study (with the exception of Alcohol Abuse)
* Report of psychotic disorder in a 1º relative
* Prenatal exposure to alcohol (mother reported to drink 3 or more drinks on an occasion or more than 3 times per month during pregnancy
* Not speaking English fluently or being a non-native English speaker, or being educated in a primary language other than English >grade 1
* Mental retardation (Full Scale IQ<70)
* Traumatic brain injury with loss of consciousness > 30 minutes or concussion in last 30 days
* Presence or history of any medical/neurologic illness that may affect brain physiology (e.g., epilepsy, Multiple Sclerosis), including focal brain lesion seen on structural MRI (all structural scans are read by a licensed radiologist)
* Current pregnancy (all females will be tested with urine screens on the day of MRI)
* Any positive alcohol screen will result in exclusion
* Inability to comprehend the consent form appropriately
* Other specific fMRI exclusions include metal devices, clips or fragments in body (orbital x-ray performed if needed)
* Female participants under 125 pounds will be excluded from participating due to the strength and side effects in this segment of the population.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2011-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey D Pearlson, MD, Principal Investigator — Yale University
Locations (1):
- Olin Neuropsychiatry Research Center at the Institute of Living, Hartford Hospital, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 82 participants were screened for eligibility and then were consented at the Olin Research Center. However, after consent and prior to group randomization, 11 participants were excluded from the study due to follow-up eligibility paperwork (i.e. psychiatric interview, family history review, etc.) for a total of 71 randomized.
Groups:
- Family History Negative (FHN): Memantine, Then Placebo: Participants received 2-20mg tablets of Memantine on the morning of the first study visit, then received 2 matching placebo tablets on the morning of the second study visit. Visits were approximately 1 week to 1 month a part on average.
  Family History Negative (FHN): People who have no affected first- or second-degree relatives.
- Family History Negative (FHN): Placebo, Then Memantine: Participants received 2 matching placebo tablets on the morning of the first study visit, then received 2-20mg tablets of Memantine on the morning of the second study visit. Visits were approximately 1 week to 1 month a part on average.
  Family History Negative (FHN): People who have no affected first- or second-degree relatives.
- Family History Positive (FHP): Memantine, Then Placebo: Participants received 2-20mg tablets of Memantine on the morning of the first study visit, then received 2 matching placebo tablets on the morning of the second study visit. Visits were approximately 1 week to 1 month a part on average.
  Family History Positive (FHP): People who have a biological father with alcoholism and at least one other first- or second-degree relative with alcoholism.
- Family History Positive (FHP): Placebo, Then Memantine: Participants received 2 matching placebo tablets on the morning of the first study visit, then received 2-20mg tablets of Memantine on the morning of the second study visit. Visits were approximately 1 week to 1 month a part on average.
  Family History Positive (FHP): People who have a biological father with alcoholism and at least one other first- or second-degree relative with alcoholism.
Period: Overall Study
Arm/Group | Family History Negative (FHN): Memantine, Then Placebo | Family History Negative (FHN): Placebo, Then Memantine | Family History Positive (FHP): Memantine, Then Placebo | Family History Positive (FHP): Placebo, Then Memantine
Started | 18 | 18 | 16 | 19
Completed | 15 | 17 | 15 | 18
Not Completed | 3 | 1 | 1 | 1
Not completed — Lost to Follow-up | 3 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Family History Positive (FHP): People who have a biological father with alcoholism and at least one other first- or second-degree relative with alcoholism.
- Family History Negative (FHN): People who have no affected first- or second-degree relatives.
- Total: Total of all reporting groups
Arm/Group | Family History Positive (FHP) | Family History Negative (FHN) | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 36 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: The number of participants analyzed is different from the overall baseline participants because a total of 6 participants (2 FHP, 4 FHN) did not complete both of the interventions (memantine, placebo) due to lost to follow-up.
  years
    number analyzed (Participants) | 33 | 32 | 65
    (all) | 24.70 [18 to 34] | 22.09 [19 to 27] | 23.42 [18 to 34]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number of participants analyzed is different from the overall baseline participants because a total of 6 participants (2 FHP, 4 FHN) did not complete both of the interventions (memantine, placebo) due to lost to follow-up.
  Participants
    number analyzed (Participants) | 33 | 32 | 65
    Female | 28 | 20 | 48
    Male | 5 | 12 | 17
Region of Enrollment [Number; unit: participants] — Population: The number of participants analyzed is different from the overall baseline participants because a total of 6 participants (2 FHP, 4 FHN) did not complete both of the interventions (memantine, placebo) due to lost to follow-up.
  participants
    United States: number analyzed (Participants) | 33 | 32 | 65
    United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Oxygenation Level Dependent (BOLD) Activation in the Amygdala During "Win" Monetary Incentive Delay (MID) Task Between Placebo and Study Medication
Description: All participants completed the fMRI Monetary Incentive Delay task on each study day. During the task, participants needed to select the correct response during "win" and "lose" conditions by pressing a button on a button box in the MRI. Participant's BOLD activation response (A measurement of oxygen level that is released to neurons since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen to perform the tasks.) was measured while they performed the task in MRI scanner.
Time Frame: 4 hours post intervention on each study day, separated by 1 week to 1 month
Population: The number of subjects analyzed differs from the overall number of subjects because analyses for this measure occurred about 48 months into recruitment.
Measure: Mean (Standard Deviation); unit: voxel wise BOLD signal
Groups:
- FHN - Memantine; FHN - Placebo: Family History Negative (FHN): People who have no affected first- or second-degree relatives.
- FHP - Memantine; FHP - Placebo: Family History Positive (FHP): People who have a biological father with alcoholism and at least one other first- or second-degree relative with alcoholism.
Arm/Group | FHN - Memantine | FHN - Placebo | FHP - Memantine | FHP - Placebo
Number analyzed (Participants) | 27 | 27 | 12 | 12
voxel wise BOLD signal | -0.6994 (3.8049) | 1.7115 (3.9355) | 0.3683 (3.9475) | 4.0298 (5.6935)
Statistical Analysis 1: Comparison: FHN - Memantine vs FHN - Placebo; Test type: Other; p = 0.032, t-test, 2 sided — P value was adjusted for multiple comparisons using FWE (family wise error) correction; A Paired t-test was performed to explore the difference between two groups; Mean Difference (Net) = 2.4109 — FHN was found to have lower mean BOLD activation while given drug compared to placebo in amygdala
Statistical Analysis 2: Comparison: FHP - Memantine vs FHP - Placebo; Test type: Other; p = 0.125, t-test, 2 sided; Median Difference (Net) = 3.6615

2. Secondary Outcome: Change in Impulsive Behavior as Measured on the Balloon Analog Risk Task (BART) Computerized Task Between Placebo and Study Medication
Description: All participants completed the BART task approximately 3 hours post drug administration on both study visits. Study days were approximately 1 week to 1 month a part. BART is a computer decision-making task that measures risk taking. Participants are presented with a series of "balloons." The object is to earn as much money as possible by pumping the balloon without popping it. The point of explosion varies from trial to trial and costs participants the money they have earned in that trial.
Time Frame: 3 hours post intervention on each study day, separated by 1 week to 1 month
Population: Participants with a family history of alcoholism (family history positive) and without a history of alcoholism (family history negative) who completed BART task.
Measure: Mean (Standard Deviation); unit: total pumps
Arm/Group | FHN - Memantine | FHN - Placebo | FHP - Memantine | FHP - Placebo
Number analyzed (Participants) | 18 | 19 | 19 | 26
total pumps | -0.12839 (1.001) | -0.04331 (1.033) | 0.2727 (0.910) | -0.0789 (1.022)

3. Secondary Outcome: Change in Impulsive Behavior as Measured on the Experimental Discounting Delay (EDT) Computerized Task Between Placebo and Study Medication
Description: All participants completed the EDT task approximately 3 hours post drug administration on both study visits. Study days were approximately 1 week to 1 month a part. EDT is a delay-discounting task that exposes participants to choice consequences during test administration. The EDT involves multiple blocks of choices, one for each delay. Choices are made between a standard amount that is delivered immediately and is certain and a probable amount that is delayed and uncertain.
Time Frame: 3 hours post intervention on each study day, separated by 1 week to 1 month
Measure: Mean (Standard Deviation); unit: responses
Arm/Group | FHN - Memantine | FHN - Placebo | FHP - Memantine | FHP - Placebo
Number analyzed (Participants) | 32 | 32 | 33 | 33
responses
  # of times "delayed" pressed in Delay Condition | 13.58831 (6.838454) | 14.13 (7.414) | 15.41029 (8.256729) | 13.64 (7.504)
  # of times "immediate" pressed in Delay Condition | 10.85871 (6.972910) | 11.84 (7.133) | 10.34057 (5.995089) | 10.22 (5.873)
  # of times "delayed" pressed in Immediate Cond. | 11.44094 (3.890267) | 11.94 (4.096) | 11.77072 (4.882568) | 11.50 (4.159)
  # of times "immediate" pressed in Immediate Cond. | 18.57818 (12.316437) | 17.74 (10.847) | 14.82459 (9.884165) | 14.39 (10.431)

4. Primary Outcome: Change in Blood Oxygenation Level Dependent (BOLD) Activation in Anterior Cingulate Cortex During "Loss" Condition of Monetary Incentive Delay (MID) Task Between Placebo and Study Medication
Description: as for outcome 1
Time Frame: 4 hours post intervention on each study day, separated by 1 week to 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: voxel wise BOLD signal
Arm/Group | FHN - Memantine | FHN - Placebo | FHP - Memantine | FHP - Placebo
Number analyzed (Participants) | 27 | 27 | 12 | 12
voxel wise BOLD signal | -0.5980 (2.9465) | 1.2368 (2.8177) | .7498 (3.1314) | 3.4762 (2.3169)
Statistical Analysis 1: Comparison: FHP - Memantine vs FHP - Placebo; Test type: Other; p = 0.356, t-test, 2 sided — P value was adjusted for multiple comparisons using FWE (family wise error) correction; Mean Difference (Net) = 2.7264 — FHP was found to have lower mean BOLD activation while given drug compared to placebo in anterior cingulate cortex
Statistical Analysis 2: Comparison: FHN - Memantine vs FHN - Placebo; Test type: Other; p = 0.009, t-test, 2 sided; Median Difference (Net) = 1.8348

ADVERSE EVENTS:
Time Frame: AE data were collected over the duration of the study (4 years).
Description: All AE information that were collected were expected side effects of the study medication.
Arm/Group | Family History Positive (FHP) | Family History Negative (FHN)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 24/35 | 26/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family History Positive (FHP) (N=35) | Family History Negative (FHN) (N=36)
Dizziness (General disorders) | 14 (14) | 12 (12)
Lightheaded (General disorders) | 19 (19) | 17 (17)
"Drunk" or "Tipsy" (General disorders) | 5 (5) | 2 (2) — Study intervention did not involve use of alcohol, however one common side effect of the study medication includes feeling "drunk."
Nausea (General disorders) | 2 (2) | 2 (2)
Vomit (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No